CLINICAL TRIAL: NCT00935584
Title: Patient Centered Evaluation of Computerized Patient Records System
Acronym: PACECPRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 07-196
Record Dates: First submitted 2009-07-07; First posted 2009-07-09 (Estimated); Results first posted 2015-11-06 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-10

CONDITIONS: Electronic Medical Records
Keywords: Communication; Doctor-patient relations; medical informatics; patient-centered care; medical records systems, computerized
MeSH Terms: conditions — Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PACE Study (Other): The study utilized a quasi-experimental pre-post intervention design. The intervention provided was physician education to improve EMR use and communication.
  Physician training in patient-centered EMR use was developed. The conceptual model of "patient-centered communication" will provide the underlying framework for the training aimed at improving physicians interviewing and communication skills.
  Interventions: Behavioral: Physician training in patient-centered emr use

INTERVENTIONS:
Behavioral: Physician training in patient-centered emr use — This intervention was performed in between the pre-intervention (Baseline) clinic visit and post intervention clinic visit.
  Other Names: Educational Workshop

SUMMARY:
The VHA is a leader in electronic medical records (EMR) use for patient care. It is believed that EMR use by doctors will improve patient-centeredness of visits, and improve clinical care. The proposed study will determine how doctors should use the EMR during patient consultations. We will also develop a training program to improve doctors ability to communicate with patients while using EMR.

DETAILED DESCRIPTION:
Anticipated Impact on Veterans Healthcare: Health information technology (HIT), including electronic medical records (EMR) has the potential to improve the quality and safety of ambulatory care. The VHA is a leader in EMR implementation. It is believed that EMR use by physicians will improve patient-centeredness of visits, and healthcare outcomes. The proposed clinical trial addresses the need for rigorous research on EMR use, patient-centered care, and relevant health outcomes. Both physician-patient communication and EMR use are cross-cutting clinical issues with broad implications for patient care within the VHA. Consequently, the proposed project is directly related to the VHA's mission to use HIT to improve the quality health care for veteran patients.

BACKGROUND/RATIONALE EMRs can potentially improve quality and safety of ambulatory care. However, little research systematically documents the effect of EMRs on patient-centered care. Studies of the EMR's effect on patient-provider communication have been observational and had small sample sizes. Overall, these studies reported varied success regarding providers integrating the EMR into office visits, and suggest that further research is needed to evaluate the effectiveness of training providers in patient-centered communication and EMR use.

OBJECTIVES The PACE aims were to study how EMR use affects patient-provider communication behaviors, and patient-centered care and related health outcomes; to develop a unique provider training program tailored to patient-centered EMR use; and to evaluate the effect of the training intervention on patient-provider communication, patient-centered care, and provider EMR use.

METHODS

The study used a quasi-experimental (pre-post intervention design) carried out in three phases:

1. Pre-intervention: A pre-intervention patient-provider visit was conducted for each patient-provider pair. Visits were video recorded and reviewed for verbal and nonverbal patient-provider communication. MORAE software was used to record provider-EMR interaction data, including page views, navigation, and mouse clicks. Data were collected for related outcomes (patient and provider satisfaction).
2. Training: Findings from pre-intervention data guided development of a multifaceted provider training intervention promoting patient-centered EMR appropriation. The training intervention was delivered via a full day training workshop and individual feedback sessions.
3. Post-intervention: A second round of visits was conducted with the same patient-provider pairs and similar data were collected as in pre-intervention. Within group analyses (pre-post) were used to test whether the training intervention resulted in significant improvements in (a) patient-centered EMR use and (b) related outcomes (patient and provider satisfaction).

IMPACT PACE findings emphasize the need to address EMR usability by the VHA hi2 (Health Informatics Initiative) and iEHR team.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age>18) male and female patients from participating study providers' practices who have an established a doctor-patient relationship with their provider and require a minimum of 2 primary care clinic visits/year based on historical clinic data.

Exclusion Criteria:

* Patients with significant communication disability (severe speech and hearing impairment, severe dementia, or a mental health condition resulting in a non-communicative patient);
* patients are considered mentally incompetent to provide informed written consent;
* a life expectancy of less than 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2010-05; Primary Completion 2013-02 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zia Agha, MD MS, Principal Investigator — VA San Diego Healthcare System, San Diego
Locations (1):
- VA San Diego Healthcare System, San Diego, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study recruited 23 primary care providers from VA San Diego and its community based outpatient clinics. For each provider we enrolled approximately 6 patients from their out-patient practice. A total of 23 physicians and 126 patients were included in the final analysis.
Groups:
- PACE Study Patients: The proposed study will use a quasi-experimental (pre-post intervention design). Pre-intervention phase consisted of baseline data collection on EMR usage and patient-physician communication.
  126 patients started the study and 77 completed the study.
- PACE Study Providers: 23 primary care providers started and 19 completed the study. 22 primary care providers participated in the educational workshop.
Period: Overall Study
Arm/Group | PACE Study Patients | PACE Study Providers
Started | 126 (Out of 128 participants consented, 2 patients had no data collected, as the clinic was cancelled.) | 23
Completed | 77 | 19
Not Completed | 49 | 4
Not completed — Withdrawal by Subject | 9 | 0
Not completed — Death | 3 | 0
Not completed — Lost to Follow-up | 8 | 0
Not completed — No show | 9 | 0
Not completed — Relocated | 3 | 0
Not completed — Patient changed provider | 3 | 0
Not completed — Provider dropped out of study | 14 | 4

BASELINE CHARACTERISTICS:
Population: Our primary analysis is based on 126 patients/clinic visits (Of the 128 visits, 2 visits had no data). The total number of enrollments were 151 (128 patients + 23 providers).
Groups:
- PACE Study Patients: The proposed study will use a quasi-experimental (pre-post intervention design) carried out in three phases.
  Physician training in patient-centered emr use: physician training in patient-centered EMR use (PACE) will be developed. The conceptual model of "patient-centered communication" will provide the underlying framework for the training aimed at improving physicians interviewing and communication skills.
- PACE Study Providers: 23 providers participated in the study. However, final analysis was based on 126 clinic visits.
- Total: Total of all reporting groups
Arm/Group | PACE Study Patients | PACE Study Providers | Total
Number analyzed (Participants) | 126 | 23 | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (13.4) | NA (NA) — Only provider gender and location was recorded. | NA (NA) — Only provider gender and location was recorded.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 17 | 21
  Male | 122 | 6 | 128
Region of Enrollment [Number; unit: participants]
  United States | 126 | 23 | 149

OUTCOME MEASURES:

1. Primary Outcome: Change in Patient's Satisfaction, Change in Provider's Satisfaction (Mean/SD)
Description: Three patient satisfaction subscales were analyzed (range 1-5 for all subscales, 1=not satisfied at all, 5=very satisfied). Subscale 1 measures physician's use of patient center communication; Subscale 2 measures clinical competence and skills; Subscale 3 measures physician interpersonal skills. Four provider satisfaction subscales were analyzed (range 1-5 for all subscales, 1=not satisfied at all, 5=very satisfied). Subscale 1 measures quality of physician-patient relation; Subscale 2 measures patient's non-demanding co-operative nature, Subscale 3 measures satisfaction with data collection; Subscale 4 measures satisfaction with use of visit time.
  Change in patient's satisfaction and change in provider's satisfaction from pre to post-intervention clinic visit was reported for the above subscales. Higher change score indicates better outcome. Mean and standard deviation were reported.
Time Frame: Baseline clinic visit and post-intervention clinic visit (over a period of 1 year)
Population: Wilcoxon signed rank test was used to analyzed the subjects using complete data (ranges from 63 to 73 for the outcomes reported below) only and mixed model method was used to analyze the subjects (ranges from 108 to126) using all available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- PACE Study: The proposed study will use a quasi-experimental (pre-post intervention design) carried out in three phases.
  Physician training in patient-centered emr use: physician training in patient-centered EMR use (PACE) will be developed. The conceptual model of "patient-centered communication" will provide the underlying framework for the training aimed at improving physicians interviewing and communication skills.
Arm/Group | PACE Study
Number analyzed (Participants) | 126
units on a scale
  Patient satisfaction/visit | -0.033 (0.454)
  Patient satisfacton/clinical skill | 0.032 (0.69)
  Patient satisfaction/interpersonal skill | -0.018 (0.386)
  Provider satisfaction/physician-patient relation | 0.077 (0.538)
  Provider satisfaction/patient's cooperation | 0.0101 (0.869)
  Provider satisfaction/data collection | 0.095 (0.686)
  Provider satisfaction/use of time | -0.035 (0.827)
Statistical Analysis 1: Comparison: PACE Study; The null hypothesis states that there is no significant change in outcome from pre-intervention clinical visit (baseline) to post-intervention clinic visit; Test type: Superiority or Other; p > 0.05, Mixed Models Analysis
Statistical Analysis 2: Comparison: PACE Study; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p > 0.05, Wilcoxon signed rank test

2. Primary Outcome: Change in Patient's Satisfaction, Change in Provider's Satisfaction (Median/Range)
Description: Three patient satisfaction subscales were analyzed (range 1-5 for all subscales, 1=not satisfied at all, 5=very satisfied). Subscale 1 measures physician's use of patient center communication; Subscale 2 measures clinical competence and skills; Subscale 3 measures physician interpersonal skills. Four provider satisfaction subscales were analyzed (range 1-5 for all subscales, 1=not satisfied at all, 5=very satisfied). Subscale 1 measures quality of physician-patient relation; Subscale 2 measures patient's non-demanding co-operative nature, Subscale 3 measures satisfaction with data collection; Subscale 4 measures satisfaction with use of visit time.
  Change in patient's satisfaction and change in provider's satisfaction from pre to post-intervention clinic visit was reported for the above subscales. Higher change score indicates better outcome. Median and range were reported.
Time Frame: Baseline clinic visit and post-intervention clinic visit (over a period of 1 year)
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | PACE Study
Number analyzed (Participants) | 126
units on a scale
  Patient satisfaction/visit | 0 [-1.44 to 1.38]
  Patient satisfaction/clinic skill | 0 [-2.33 to 3.33]
  Patient satisfaction/interpersonal skill | 0 [-2 to 1.33]
  Provider satisfaction/physician-patient relation | 0 [-1.75 to 2]
  Provider satisfaction/patient's cooperation | 0 [-1.67 to 3]
  Provider satisfaction/data collection | 0 [-1.67 to 2]
  Provider satisfaction/use of time | 0 [-3 to 1.67]
Statistical Analysis 1: Comparison: PACE Study; The null hypothesis is that there is no significant change in outcome from pre to post visit; Test type: Superiority or Other; p > 0.05, Mixed Models Analysis
Statistical Analysis 2: Comparison: PACE Study; The null hypothesis is that there is no significant change in outcome from pre to post visit; Test type: Superiority or Other; p > 0.05, Wicoxon signed rank test

3. Primary Outcome: Change in Patient Engagement
Description: Change in proportion of time spent on physician-patient communication from pre to post-intervention clinic visit was calculated. Positive change indicates increased time spent on patient communication. Mean and standard deviation of outcomes were reported in this table.
Time Frame: Baseline clinic visit and post-intervention clinic visit (over a period of 1 year)
Population: Wilcoxon signed rank test was used to analyzed the subjects using complete data (n=72 for the outcomes reported below) only and mixed model method was used to analyze the subjects (n=125) using all available data.
Measure: Mean (Standard Deviation); unit: percentage of total visit time
Arm/Group | PACE Study
Number analyzed (Participants) | 125
percentage of total visit time
  Time spent on patient and companion | 2.9 (15.2)
  Time spent on physical exam | -1.4 (14.7)
  Time spent on EMR | -1.6 (16.6)
Statistical Analysis 1: Comparison: PACE Study; The null hypothesis is that there is no significant change in patient engagement from pre to post visit; Test type: Superiority or Other; p > 0.05, Mixed Models Analysis
Statistical Analysis 2: Comparison: PACE Study; The null hypothesis is that there is no significant change in patient engagement from pre to post visit; Test type: Superiority or Other; p > 0.05, Wilcoxon signed rank test

4. Primary Outcome: Change in Total Number of EMR Mouse Click Per Visit (Mean/SD)
Description: For EMR use, we assessed the change in total number of mouse click per-visit, positive score indicates increased EMR use. Mean and standard deviation of outcome were reported in this table.
Time Frame: Baseline clinic visit and post-intervention clinic visit (over a period of 1 year)
Population: Wilcoxon signed rank test was used to analyzed the subjects using complete data (n= 60 for the outcomes reported below) only and mixed model method was used to analyze the subjects (n=119) using all available data.
Measure: Mean (Standard Deviation); unit: EMR mouse clicks per visit
Arm/Group | PACE Study
Number analyzed (Participants) | 126
EMR mouse clicks per visit | -1.22 (155)
Statistical Analysis 1: Comparison: PACE Study; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis
Statistical Analysis 2: Comparison: PACE Study; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, Wilcoxon signed rank test

5. Primary Outcome: Change in Total Number of EMR Mouse Click Per Visit (Median/Range)
Description: For EMR use, we assessed the change in total number of mouse click per-visit, positive score indicates increased EMR use.
Time Frame: Baseline clinic visit and post-intervention clinic visit (over a period of 1 year)
Population: Wilcoxon signed rank test was used to analyzed the subjects using complete data (n=60 for the outcomes reported below) only and mixed model method was used to analyze the subjects (n=119) using all available data.
Measure: Median (Full Range); unit: EMR mouse clicks per visit
Arm/Group | PACE Study
Number analyzed (Participants) | 126
EMR mouse clicks per visit | -2 [-412 to 303]
Statistical Analysis 1: Comparison: PACE Study; The null hypothesis is that there is no significant change in outcome from pre to post visit; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis
Statistical Analysis 2: Comparison: PACE Study; The null hypothesis is that there is no significant change in outcome from pre to post visit; Test type: Superiority or Other; p < 0.05, Wilcoxon signed rank test

6. Primary Outcome: Change in EMR Mouse Click Per Minute Per Visit (Mean/SD)
Time Frame: Baseline clinic visit and post-intervention clinic visit (over a period of 1 year)
Population: Wilcoxon signed rank test was used to analyzed the subjects using complete data (n=56 for the outcomes reported below) only and mixed model method was used to analyze the subjects (n=119) using all available data.
Measure: Mean (Standard Deviation); unit: EMR mouse clicks per minute per visit
Arm/Group | PACE Study
Number analyzed (Participants) | 126
EMR mouse clicks per minute per visit | -0.089 (3.11)
Statistical Analysis 1: Comparison: PACE Study; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis
Statistical Analysis 2: Comparison: PACE Study; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, Wilcoxon signed rank test

7. Primary Outcome: Change in EMR Mouse Click Per Minute Per Visit (Median/Range)
Description: For EMR use, we assessed the change in the average number of mouse clicks per minute per-visit, positive score indicates increased EMR use.
Time Frame: Baseline clinic visit and post-intervention clinic visit (over a period of 1 year)
Population: as for outcome 6
Measure: Median (Full Range); unit: EMR mouse clicks per minute per visit
Arm/Group | PACE Study
Number analyzed (Participants) | 126
EMR mouse clicks per minute per visit | 0.005 [-7.13 to 5.84]

ADVERSE EVENTS:
Description: Adverse events were not expected, therefore not collected for providers and patients.
  Threshold for adverse event was reported as 0 for technical purpose (the system does not allow us to save if not entering).
Arm/Group | PACE Study
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Study limitations include inability to capture EHR activity outside the visit, study only primary care providers at a single organization (VA) and only one EHR system, this limits generalizability of the findings to other setting.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No